CLINICAL TRIAL: NCT00670124
Title: Pilot Trial on the Effect of Mild Hypothermia on Intracranial Pressure in Patients With Hyperacute Liver Failure
Brief Title: Hypothermia to Prevent High Intracranial Pressure in Patients With Acute Liver Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: University Hospital Birmingham (Other); Northwestern University Feinberg School of Medicine (Other)
Responsible Party: Principal Investigator, Dr. Fin Stolze Larsen, Head of Research Unit, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALFHypothermia01
Record Dates: First submitted 2008-04-29; First posted 2008-05-01 (Estimated); Last update posted 2014-11-05 (Estimated); Status verified 2014-11

CONDITIONS: Acute Liver Failure; Intracranial Hypertension
MeSH Terms: conditions — Liver Failure, Acute; Intracranial Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (No Intervention): Standard medical treatment
- 2 (Active Comparator): Standard medical treatment plus hypothermia (33°C) maintained for 72 hours
  Interventions: Device: Hypothermia by the use of Blanketrol II, Cincinnati Sub-Zero

INTERVENTIONS:
Device: Hypothermia by the use of Blanketrol II, Cincinnati Sub-Zero — The patients are placed on a cooling mattress and body-core temperature is regulated to 33° C.
  Other Names: Cooling device: Blanketrol II, Cincinnati Sub-Zero
  Arms: 2

SUMMARY:
Treatment options in patients with high intracranial pressure due to acute liver failure are limited. This study intends to evaluate the effect of prophylactic hypothermia on preventing high intracranial pressure and compromised cerebral oxidative metabolism.

DETAILED DESCRIPTION:
Acute liver failure (ALF) is associated with a high mortality. With severe hepatic encephalopathy and elevated arterial ammonia concentration (< 200 micromol/L) more than 50% of the patients will develop high intracranial pressure (ICP) and risk cerebral incarceration and death. The therapeutic options are limited in treating and preventing this condition and new interventions are much sought after. As in hypothermia used for patients after cardiac resuscitation it could be speculated that hypothermia and the reduced cerebral metabolic rate would contribute to neuroprotection and reduce the risk of cerebral hypertension in patients with ALF. We have designed this open, randomized and unblinded study in order to evaluate the effect of prophylactic hypothermia on ICP, cerebral hemodynamics and oxidative metabolism. Patients are randomized to standard medical treatment (SMT) or SMT and hypothermia 33° C for 72 hours using a cooling mattress (Blanketrol II, Cincinnati Sub-Zero). All patients will receive mechanical ventilation, antibiotics, inotropic support and monitored with invasive and non-invasive equipment in accordance to local guidelines. In Copenhagen monitoring cerebral hemodynamics includes:

Placement of a intracranial pressure measuring catheter (Camino (R), Integra) for monitoring ICP. Furthermore, a microdialysis catheter (CMA-70) placed in brain cortex is used for monitoring brain metabolism. Finally, cerebral perfusion can be monitored by measuring mean flow velocity using transcranial doppler and/or oxygen saturation in blood from the jugular vein.

Ethical considerations:

The Helsinki II declaration will be followed and informed consent is mandatory for enrollment. In any patient where hypothermia is believed or suspected to be harmful the study should be stopped and the primary investigator should be notified immediately. All adverse effects will be recorded and published together with the full paper.

ELIGIBILITY:
Inclusion Criteria:

* acute liver failure
* and hepatic encephalopathy stage 3 or 4
* and informed and written consent by closest relative(s)
* and arterial ammonia concentration above 150 micromol/L or clinical suspicion of cerebral edema
* and an ICP-measuring device

Exclusion Criteria:

* no or withdrawn informed consent
* pregnant or breast feeding women
* uncontrollable infection
* hemodynamically instable patients
* active bleeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2005-01; Primary Completion 2011-01 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
The effect of hypothermia on preventing development of ICP higher than 25 mmHg | 72 hours

SECONDARY OUTCOMES:
The effect of hypothermia on preserving normal cerebral oxidative metabolism evaluated by cerebral microdialysis | 72 hours
The effect of hypothermia on severity of infections | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Fin S Larsen, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (4):
- Division of Hepatology, Feinberg School of Medicine, Northwestern University, Chicago, Illinois, United States
- Department of hepatology, Rigshospitalet, Copenhagen, Denmark
- United Kingdom (2):
  - Dept. of Intensive Care, Birmingham
  - Institute for Liver Studies, King's College Hospital, London